CLINICAL TRIAL: NCT04103268
Title: Neutrophil Phenotypic Profiling and Organ Injury Assessment in Patients With Sepsis
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00031930
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis
  Interventions: Other: sepsis
- Control

INTERVENTIONS:
Other: sepsis — patients in the ICU with infection called sepsis
  Groups: Sepsis

SUMMARY:
In this research study we want to learn more about the character of neutrophils that are present in the blood of children with sepsis. Sepsis is a severe type of infection, affecting various parts of the body. Neutrophils are a type of white blood cell that are part of the body's immune system. Even though neutrophils are important in getting rid of germs, they also may be harmful to parts of the body by causing injury in organs in patients with sepsis. Neutrophils can change their character in sepsis. Because of this, it is important for doctors to know what kind of neutrophils are in the blood of children with sepsis so that they can work to develop therapies to prevent these cells from being harmful.

ELIGIBILITY:
Inclusion criteria Patients will be eligible for enrollment as septic patients if they

* Are < 18 years old
* Meet the definition of sepsis described in the study design section above. Patients will be eligible for enrollment as control patients if they
* Are < 18 years old
* Are scheduled for an elective surgical procedure and need preoperative blood draw or will have an intravenous catheter placed for the purpose of their surgical procedure.

Exclusion criteria Patients will be ineligible for enrollment in either control or sepsis group if any of the followings is present or anticipated

* Congenital cardiac disease
* On chronic immunosuppressive drugs such as chronic corticosteroid use, or preexisting immunodeficiency diseases

Ages: 1 Month to 17 Years | Sex: All
Age Groups: Child
Study Population: We will enroll pediatric patients with sepsis in an ICU at Boston Children's Hospital and patients without sepsis presenting for an elective surgical procedure at Boston Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
neutrophil populations | up to 1 month
  compare gene expression in neutrophils between sepsis patients and non-sepsis patients in pediatric population to report unregulated and down regulated genes

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Yuki, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Alhamdan F, Gianoli S, Yuki K, Koutsogiannaki S. Single-cell analysis of B cell dysregulation in pediatric sepsis stratified by disease severity. Sci Rep. 2025 Dec 31;16(1):3987. doi: 10.1038/s41598-025-34126-9. PMID 41476192